CLINICAL TRIAL: NCT01031056
Title: Collection of Biospecimen and Clinical Information in Patients With Gastrointestinal Cancers
Brief Title: Collection of Biospecimen & Clinical Information in Patients w/ Gastrointestinal Cancers
Status: Withdrawn | Type: Observational
Why Stopped: Change in research focus
Sponsor: Stanford University (Other)
Collaborators: Caring for Carcinoid Foundation (Other); GI Cancer Research Gift Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: SU-09092009-3840; GI0004
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Gastrointestinal Neoplasms; Gynecologic Cancers; Gynecologic Cancers Cervical Cancer; Gastric (Stomach) Cancer; Gastro-Esophageal(GE) Junction Cancer; Gastrointenstinal Stromal Tumor (GIST); Colon/Rectal Cancer; Colon/Rectal Cancer Colon Cancer; Colon/Rectal Cancer Rectal Cancer; Colon/Rectal Cancer Anal Cancer; Anal Cancer; Hepatobiliary Cancers; Hepatobiliary Cancers Liver; Pancreatic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study requires that we obtain archived tumor and normal tissue and blood.

INTERVENTIONS:
Procedure: Blood Draw
Procedure: Frozen Tumor Specimens

SUMMARY:
We have an active research program in gastrointestinal cancers including clinical trials, epidemiologic, and translational studies. We would like to establish a biospecimen bank linked to useful clinical information in order to learn more about diagnostic, predictive and prognostic markers for gastrointestinal cancers.

PRIMARY OBJECTIVES:

1. To collect and store tumor and normal tissue (previously collected paraffin embedded or frozen specimen) and blood in patients with gastrointestinal (GI) cancers.

SECONDARY OBJECTIVES:

1. Collect detailed clinical information via a patient questionnaire that includes demographic, socioeconomic, lifestyle, family, past medical, medication and cancer histories
2. Collect details about the tumor specimen extracted from patient charts.

ELIGIBILITY:
Inclusion Criteria:1. Patients are eligible if they have a histologically proven gastrointestinal cancer (esophageal, gastroesophageal junction, gastric, small intestine, appendix, colon, rectum, anus, liver, gallbladder, bile ducts, pancreas, neuroendocrine, and GI stromal tumor).

2. 18 years of age or older

3. Ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
None: Biospecimen will be collected for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Teri A Longacre M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States